CLINICAL TRIAL: NCT05267782
Title: Correlation Between New O3 Regional Oximetry, Electroencephalography and the Somatosensory Evoked Potential in Carotid Endarterectomy Surgery
Status: Recruiting | Type: Observational
Sponsor: Cleveland Clinic Abu Dhabi (Other)
Responsible Party: Principal Investigator, Boris Tufegdzic, Associate Professor, Cleveland Clinic Abu Dhabi
Other Study IDs: A-2022-005
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Carotid Endarterectomy
Keywords: O3 regional oximetry; somatosensory evoked potential; electroencephalography; carotid endarterectomy surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Masimo's O3 Regional Oximetry — Correlation between new O3 regional oximetry monitoring, electroencephalography and somatosensory evoked potential in carotid endarterectomy and data collection during different stages of anaesthesia and correlation with new O3 regional oximetry

SUMMARY:
Carotid endarterectomy (CEA) is one of the modalities to treat carotid artery disease. One of the perioperative complications of this surgery includes stroke, a condition that occurs when the blood supply to part of your brain is interrupted or reduced. To prevent cerebral ischemia during carotid endarterectomy several methods have been employed in clinical practice, such as awake neurocognitive assessment, electroencephalography, evoked potentials, transcranial Doppler, carotid stump pressure, and near infrared spectroscopy (Regional Oximetry).

Meta-analysis published by Nwachuku EL and colleagues suggests that intraoperative somatosensory evoked potential (SSEP) is a highly specific test in predicting neurological outcome following CEA. Sridharan and colleagues advise multimodality in intraoperative monitoring, with simultaneous use of EEG and SSEP which will improve the diagnostic accuracy. Use of regional oximetry as a continuous, real time and non-invasive monitoring, during CEA is controversial, with pros and cons studies that do not contribute to a clear picture of its application in everyday clinical practice.

Masimo's O3 Regional Oximetry is new monitoring approved in 2020 by FDA for monitoring somatic tissue oxygenation saturation in all patient populations and for monitoring relative changes in haemoglobin, oxyhaemoglobin, and deoxyhaemoglobin in adult brains. This monitoring can help clinicians to monitor cerebral oxygenation in situations in which pulse oximetry alone may not be fully indicative of the oxygen in the brain. One such example is carotid endarterectomy (CEA).

Masimo's O3 regional oximetry is integrated part of the SedLine® Brain Function Monitoring (Masimo, Irvine, California, USA, 1989) on the Root® Patient Monitoring Platform. Sensors are equipped within Masimo Open Connect (MOC-9) modules which are applied to the patient's forehead and connected to the Masimo Root® patient monitoring and connectivity platform.

Masimo's O3 Regional Oximetry provides regional or tissue haemoglobin oxygen saturation and unlike peripheral pulse oximetry, which reflects the body's general arterial blood oxygenation, O3 provides information about the local tissue's haemoglobin oxygen saturation, both in cerebral and somatic applications. This information provides additional insight that may help inform clinicians of changes in cerebral or somatic tissue oxygen levels.

Regional Oximetry is already part of the standard monitoring used during CEA in Cleveland Clinic Abu Dhabi, together with electroencephalography and the somatosensory evoked potentials.

Using new Masimo's O3 regional oximetry monitoring (same sensor, only the module is new with new parameters) we will have additional parameters that have not been analysed before:

* Δbase
* ΔSpO2
* ΔcHbi
* Δ HHbi
* ΔO2Hbi

With this in mind, the authors would like to analyse the correlation between new Masimo's O3 regional oximetry parameters, EEG and SSEP in CEA.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects older than 18 years of age
2. Subjects undergoing carotid endarterectomy.
3. American Society of Anaesthesiologists Classification (ASA) score I to III.

Exclusion Criteria:

1. American Society of Anaesthesiologists Classification (ASA) score IV and V.
2. Subject has skin abnormalities affecting the sensor placement
3. Emergency cases
4. Cognitive/Mentally impaired or unable to provide consent
5. Pregnant subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is prospective observational pilot study and only 10 subjects will be recruited after application of the below inclusion/exclusion criteria. Subjects will be included only if they sign informed consent for study. The anticipated duration of subject's participation in this study will not exceed duration of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between new O3 regional oximetry monitoring, electroencephalography and SSEP in CEA. | The anticipated duration will not exceed duration of surgery.

SECONDARY OUTCOMES:
Data collection during different stages of anaesthesia and correlation with new O3 regional oximetry | The anticipated duration will not exceed duration of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Abu Dhabi, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nwachuku EL, Balzer JR, Yabes JG, Habeych ME, Crammond DJ, Thirumala PD. Diagnostic value of somatosensory evoked potential changes during carotid endarterectomy: a systematic review and meta-analysis. JAMA Neurol. 2015 Jan;72(1):73-80. doi: 10.1001/jamaneurol.2014.3071. PMID 25383418
- [Background] Domenick Sridharan N, Thirumala P, Chaer R, Balzer J, Long B, Crammond D, Makaroun M, Avgerinos E. Predictors of cross-clamp-induced intraoperative monitoring changes during carotid endarterectomy using both electroencephalography and somatosensory evoked potentials. J Vasc Surg. 2018 Jan;67(1):191-198. doi: 10.1016/j.jvs.2017.04.064. Epub 2017 Jul 5. PMID 28688529
- [Background] Friedell ML, Clark JM, Graham DA, Isley MR, Zhang XF. Cerebral oximetry does not correlate with electroencephalography and somatosensory evoked potentials in determining the need for shunting during carotid endarterectomy. J Vasc Surg. 2008 Sep;48(3):601-6. doi: 10.1016/j.jvs.2008.04.065. Epub 2008 Jul 18. PMID 18639412
- [Background] Tan TW, Garcia-Toca M, Marcaccio EJ Jr, Carney WI Jr, Machan JT, Slaiby JM. Predictors of shunt during carotid endarterectomy with routine electroencephalography monitoring. J Vasc Surg. 2009 Jun;49(6):1374-8. doi: 10.1016/j.jvs.2009.02.206. PMID 19497494
- [Background] https://www.masimo.com/technology/brain-monitoring/cerebral-oximetry
- [Background] https://www.masimo.com/siteassets/us/documents/pdf/plm_11661c_brochure_o3_series_us.pdf